CLINICAL TRIAL: NCT01551537
Title: Post-marketing Surveillance (PMS) of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) -16/18 Vaccine, Cervarix™ When Administered to Healthy Females According to the Prescribing Information in Sri Lanka
Brief Title: Post-marketing Surveillance of GSK Biologicals' Cervarix™ When Administered to Healthy Females in Sri Lanka
Status: Withdrawn | Type: Observational
Why Stopped: Lack of clarity regarding the PMS study requirement from the RA and Ethics committee hence it was concluded GSK will submit local PSURs
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113763
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Human Papillomavirus Infection
Keywords: Healthy females; Post-marketing surveillance (PMS); Human papillomavirus vaccine; Sri Lanka; Cervarix
MeSH Terms: conditions — Papillomavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort Group: Healthy females aged 10 years and above will receive 1, 2 or 3 doses of Cervarix as per the Prescribing Information (PI) in Sri Lanka.
  Interventions: Other: Cervarix data collection; Other: Data Collection

INTERVENTIONS:
Other: Cervarix data collection — Safety monitoring: recording of all AEs during the study period using diary cards, follow-up visit or telephone contact.
Other: Data Collection — All adverse events will be recorded by diary card, follow-up visit or telephone contact.

SUMMARY:
This PMS study aims to collect safety and reactogenicity data of Cervarix in the local population as per the licensing requirement of the Sri Lankan regulatory authority.

DETAILED DESCRIPTION:
Subjects who received one or two doses of Cervarix prior to the start of this PMS study can also be enrolled in the study. These subjects would receive either 2 doses or 1 dose respectively after being enrolled in the study.

Since there is lack of clarity regarding the PMS study requirement (both from Regulatory agency and Ethics Committee), it was decided that GSK will submit Local PSURs on a regular basis as desired by Local regulatory agency. The same is communicated to Regulatory agency and if they want something more they are requested to revert back with specific requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s)/ LAR(s) can and will comply with the requirements of the protocol should be enrolled in the PMS study.
* A female aged 10 years and above at the time of the first vaccination.
* Written informed consent obtained from the subject. For subjects below the legal age of consent, written informed consent must be obtained from the parent(s)/LAR(s) of the subject and informed assent must be obtained from the subject. Where subject/subject's parent(s)/LAR(s) are illiterate, the consent form will be countersigned by an impartial witness.
* Subjects of childbearing potential must not be pregnant. Absence of pregnancy should be verified as per the investigator's clinical judgement.

Exclusion Criteria:

* Subjects with contraindication according to the locally approved PI.
* Child in care.
* Previous administration of more than two doses of Cervarix.
* Previous vaccination with a HPV vaccine other than Cervarix.
* Planned administration of another HPV vaccine other than Cervarix during the PMS study.

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy females aged 10 years and above who will receive Cervarix as a part of routine practice as per the PI in Sri Lanka.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited local adverse events (AEs). | During the 7-day period (Days 0-6) following any dose of Cervarix and overall.
Occurrence of solicited general AEs. | During the 7-day period (Days 0-6) following any dose of Cervarix and overall.
Occurrence of unsolicited AEs. | During the 30-day period (Days 0-29) following any dose of Cervarix and overall.
Occurrence of any Serious adverse events (SAEs) and SAE(s) causally related to vaccination. | Throughout the PMS study period (up to six months after the last dose of Cervarix).
Occurrence of potential Immune-Mediated Diseases (pIMDs). | Throughout the PMS study period (up to six months after the last dose of Cervarix).
Occurrence of Medically Significant Condition (MSCs). | Throughout the PMS study period (up to six months after the last dose of Cervarix).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline